CLINICAL TRIAL: NCT06420492
Title: Study of Novel Therapeutics for Acute Remedy of Colitis
Acronym: SHARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua Korzenik, MD-Director, Brigham and Women's Hospital Crohn's and Colitis Center, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001885
Record Dates: First submitted 2024-05-06; First posted 2024-05-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis Chronic Moderate; Ulcerative Colitis Chronic Severe
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: This is an open-label study in which everyone will receive active treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BRS201 Arm (Experimental): In Group 1 of the study, subjects will take oral study drug at 1.2g daily, PO with 120mg oral butyrate twice daily (240mg daily) for 4 weeks.
  In Group 3 of the study, subjects will take oral study drug at 1.2g twice daily, PO (2.4g daily) with 120mg oral butyrate twice daily (240mg daily) for 4 weeks.
  In Group 3 of the study, subjects will take oral study drug at 1.2g twice daily, PO (2.4g daily) with 120mg oral butyrate twice daily (240mg daily) for 4 weeks. Subjects will also receive a one time 2.5g dose of study drug at initiation.
  In Group 4 of the study, subjects will repeat the previous conditions of the group that proves to be the most effective. Subjects in Group 4 will undergo two flexible sigmoidoscopies, one at screening and one at week 4.
  Interventions: Drug: BRS201

INTERVENTIONS:
Drug: BRS201 — Groups 1, 2, 3, and 4 will all contain 5 subjects each, with each subject receiving active study drug for four weeks.

SUMMARY:
This study is a clinical trial being done to investigate the efficacy of drug BRS201 as a treatment in patients with acute ulcerative colitis. Patients who qualify are adults who have not responded to treatments for their severe ulcerative colitis. Participation in this study will take 12 weeks long and the study is structured as an open-label pilot study in which participants will take the study drug for 4 weeks in the form of an oral medication. Participation may also involve receiving an IV dose of the medication. The study will require participants to attend 8 study visits, all of which will be conducted at a study site. Participation will involve taking an oral medication twice daily, tracking the medication in a log, and getting blood drawn and giving a stool and urine sample for a few lab tests throughout the study. Participants may also undergo a flexible sigmoidoscopy at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Severe outpatient or hospitalized for an acute UC flare
* Ability to give consent
* Patients with a confirmed diagnosis of UC for > 3 months
* History of ≥ 15 cm of colonic involvement as confirmed by colonoscopy
* Patients with primary sclerosing cholangitis are eligible to enroll
* Patients will have failed 5 days of oral prednisone 30 mg or greater for 5 days and still having a SCCAI of > 6
* Patients who are taking 20mg or less of oral prednisone and plan to stay at that dose during their participation in the study
* Accepted medications:

  * Anti-TNF agents are permissible if the patient has been taking them for at least 10 weeks and anticipates to maintain a steady for the duration of the study.
  * Rinvoq (Upadacitinib) is permissible if the subject has been taking this medication for at least 4 weeks and anticipates to maintain a steady dose for the duration of the study.
  * Xeljanz (Tofacitinib) is permissible if the subject has been taking this medication for at least 4 weeks and anticipates to maintain a steady dose for the duration of the study.
  * Other biologics are permissible if the subject has been taking the medication for at least 10 weeks and anticipates to maintain a steady dose for the duration of the study

Exclusion Criteria:

* History of uncontrolled hypertension with systolic BP > 140 and systolic BP > 90
* Chronic kidney disease as defined by GFR <55mL/min
* Impaired hepatic function (transaminases elevated > 2.5 x ULN) unless due to PSC
* Evidence of C. difficile (Negative test result within 1 month is acceptable)
* Infectious Colitis or drug induced colitis
* Crohn's Disease or Indeterminate colitis
* Decompensated liver disease
* Patients who are pregnant or breastfeeding
* Patients who have a confirmed malignancy or cancer within 5 years
* Congenital or acquired immunodeficiencies
* Other comorbidities including: Diabetes mellitus, systemic lupus
* Participation in a therapeutic clinical trial in the preceding 30 days or simultaneously during this trial
* Patients with a history or risk of cardiovascular conditions, including arrhythmia, long QT syndrome, congestive heart failure, stroke, or coronary artery disease
* Prohibited medications:

  * Rinvoq (Upadacitinib): Subjects will be excluded from this study if their last dose of this medication was administered within 4 weeks. If subjects have stopped taking this medication and their last dose was administered more than 4 weeks prior to enrollment, they will be eligible for participation.
  * Xeljanz (Tofacitinib): Subjects will be excluded from this study if their last dose of this medication was administered within 4 weeks. If subjects have stopped taking this medication and their last dose was administered more than 4 weeks prior to enrollment, they will be eligible for participation.
  * Other Medications: Subjects will be excluded from this study if they stopped taking any other medications for ulcerative colitis within 8 weeks. If subjects have stopped taking the medication and their last dose was more than 8 weeks prior to enrollment, they will be eligible for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Sulfur Metabolism | 4 weeks
  The primary measure of dose response will be urinary measures of sulfur metabolism including a > 50% reduction from pretreatment levels sulfate, and thiosulfate.

SECONDARY OUTCOMES:
Simple Clinical Colitis Activity Index (SCCAI) | 12 weeks
  Clinical symptoms assessed by SCCAI which measures patient reported outcomes on a scale of 0 to 19, where a higher score indicates more severe activity and active disease is a score of 5 or more.
Plasma nitrite, nitrate, or nitrosothiol | 8 weeks
  Correlation between changes in plasma nitrite, nitrate or nitrosothiol level in relation to calprotectin
Normalization of fecal calprotectin lab measurements | 8 weeks
  The capacity of study drug to normalize fecal calprotectin levels from baseline (week 0) compared to end of active treatment (4 weeks) and at week 6.
Reduction in fecal calprotectin lab measurements | 4 weeks
  Reduction in fecal calprotectin to < ULN at the end of active treatment
Mayo Score | 4 weeks
  The primary endpoint for this study is change in Total Mayo Score with improvement being a reduction in 3 points and remission being a score of 0 or 1 from day 0 to end of week 4 (at second flexible sigmoidoscopy).
Tissue Analysis | 4 weeks
  Analysis of tissue metabolomics and proteomics at day 0 vs day 28;
Mitochondria evaluation | 12 weeks
  Changes in mitochondria on EM evaluation
Urine Assays | 12 weeks
  Urine levels for thiosulfate, thiocyanate, nitrate and nitrite;

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States